CLINICAL TRIAL: NCT05474417
Title: The Effects of the CF Carrier State on the Kidneys and Pancreas
Status: Recruiting | Type: Observational
Sponsor: Philip Polgreen (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Philip Polgreen, Professor, Internal Medicine, University of Iowa
Organization: University of Iowa (Other)
Other Study IDs: 202012447; 5P30DK054759 (NIH)
Record Dates: First submitted 2022-07-22; First posted 2022-07-26 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Carrier State; Pancreatic Disease; Kidney Diseases
MeSH Terms: conditions — Pancreatic Diseases; Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood will be collected from all participants. Urine and/or stool samples will be collected from a subset of participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cystic Fibrosis Carrier Group: Participants who have been identified as Cystic Fibrosis Carriers via previous genetic testing.
- Control Group: Participants who have been identified as not being Cystic Fibrosis Carriers via previous genetic testing.

SUMMARY:
The overarching hypothesis is that CF carriers are at increased risk for developing most of the extrapulmonary conditions associated with CF compared to the general population. Specifically, it is hypothesized that this pilot data will detect subclinical evidence of pancreatic and kidney disorders among CF carriers. This will be determined by bringing CF carriers and controls to the CRU for one visit where they will answer survey questions and undergo laboratory testing. Additionally, they will collect urine and stool samples at home that will be sent to outside laboratories for testing.

DETAILED DESCRIPTION:
There are 2 main study components- a clinic visit (all participants) and at-home specimen collections (volunteer subsample only). Each procedure is described below.

Clinic Visit Procedures (all participants):

Height- Height will be measured to the nearest 0.5 cm. Shoes should be removed.

Weight- Weight will be measured to the nearest 0.5 kg. Shoes and any extra jackets/sweaters/layers should be removed.

Blood Pressure- Blood pressure will be measured using the following procedures- Make sure that the participant hasn't smoked for 20 minutes prior to the BP measurement. Remove all clothing that covers the location of the cuff placement. Have the participant sit comfortably in a chair, with back supported, legs uncrossed and feet flat on the floor, arm supported at the level of the heart on a table, palm facing upward. Be sure to choose a cuff that correctly fits the participant's arm size. The lower end of the cuff should be ½ to 1 inch above the inner side of the elbow joint. The middle of the cuff should be at the level of the right atrium. Place the cuff snugly around the bare upper arm so that you can only insert one finger between the cuff and the arm.

Blood Draws/2-Hour OGTT- The participant should be active and eat a regular diet for three days prior to the test. They should be instructed not to eat or drink anything except water for at least 8 hours before the test. Someone trained in phlebotomy will insert an IV into the patient's arm so that blood draws can occur before and after the oral glucose tolerance test (OGTT). They will draw 2 tubes of blood (one 3 ml lavender top tube for HbA1C and one 4.5 ml green plasma separator tube for glucose, insulin, c-peptide, and lipid values). Then, a team member will provide the participant with a chilled Fisherbrand Glucose Tolerance Test Beverage (10 oz beverage, 75 g concentration) to drink. The participant must drink the entire beverage within 5 minutes. The patient should remain seated during the 2-hours of the test. They should not eat or drink anything except for plain water during the test (no mints, cough drops, chewing gum, or smoking).

At the 1-hour mark, 1 tube of blood (4.5 ml green plasma separator tube for glucose and insulin values) will be drawn.

Once the 2 hours have passed, 2 more tubes of blood (one 3 ml lavender top tube for c-reactive protein, calprotectin, and lactoferrin and one 4.5 ml green plasma separator tube for glucose and insulin values) will be drawn.

During the downtime between blood draws, the participant will answer the questions from the baseline survey and report their current medications interview-style with the research team member.

This visit is expected to last 3-4 hours.

Home Specimen Collection (volunteer subsample only; volunteers may do urine and/or stool samples):

Participants will be given specimen collection containers and instructions on collecting the 24-hour urine sample and/or stool sample, whichever they volunteer to collect. Finally, a date, time, and meeting location will be scheduled to return the samples to the research team.

ELIGIBILITY:
CF Carrier Inclusion Criteria:

* A CF Carrier identified via genetic testing

Control Inclusion Criteria:

* No previous CF carrier test results

Exclusion Criteria:

* CF patient status
* Unable to speak English
* Currently pregnant
* Unable to provide written informed consent
* Prisoner status
* Currently taking any medications for the treatment of diabetes

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: CF Carriers and Controls who are not CF carriers.
Sampling Method: Non-Probability Sample
Enrollment: 1250 (Estimated)
Dates: Start 2021-12-20 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Comparison of Glucose Values | At baseline
  Comparison of glucose values in cystic fibrosis carrier group vs control group via t-tests.
Comparison of Insulin Values | At baseline
  Comparison of insulin values in cystic fibrosis carrier group vs control group via t-tests.

SECONDARY OUTCOMES:
Comparison of C-Reactive Protein Values | At baseline
  Comparison of c-reactive protein values in cystic fibrosis carrier group vs control group via t-tests.
Comparison of Lactoferrin Values | At baseline
  Comparison of lactoferrin values in cystic fibrosis carrier group vs control group via t-tests.
Comparison of Calprotectin Values | At baseline
  Comparison of calprotectin values in cystic fibrosis carrier group vs control group via t-tests.
Comparison of Lipid Values | At baseline
  Comparison of lipid values in cystic fibrosis carrier group vs control group via t-tests.

CONTACTS AND LOCATIONS:
Overall Officials: Philip M Polgreen, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No